CLINICAL TRIAL: NCT03981016
Title: "In Population" Study of Medical and Surgical Management of Patients With Brain Metastases
Brief Title: Medical and Surgical Management of Patients With Brain Metastases
Acronym: CEREMET-LR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICM-URC-2014/21
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Central Nervous System Tumor
Keywords: Nervous; Central; Tumor; System
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): For the patients include in the study :
  * blood samples collected at different times : Before surgery and during the post-operative visit and
  * frozen tumor samples and / or paraffin samples at the time of surgery and- paraffin around tumor samples at the time of surgery
  Interventions: Other: Biological collection

INTERVENTIONS:
Other: Biological collection — * blood samples collected at different times : Before surgery and during the post-operative visit and
  * frozen tumor samples and / or paraffin samples at the time of surgery and- paraffin around tumor samples at the time of surgery

SUMMARY:
The integrated cancer research site (SIRIC) of Montpellier proposes to develop a prospective and regional Clinical Database Project and regional biological collection (blood and tumor samples), which is an expanding data collection designed to contribute to a better understand the patient's management with brain metastases including quality of life and neuropsychological/cognitive aspects.

DETAILED DESCRIPTION:
Brain metastases (BM) represent the first cause of tumors of the central nervous system. Mortality, morbidity (cognitive disorders, neurological deficits, etc.) and their consequences on the quantity and the quality of life are very high. BM represent a real public health problem. The incidence is increasing related to the ageing of the population and the increase of cancer patient's survival rate. The medico-surgical care has highly evolved (neurosurgical progress, radiosurgery, stereotaxic radiotherapy and new chemo and targeted therapy).

Every histological or biological profile requires a specific evaluation, and management. Clinical trials are the reference to establish the efficacy and the toxicity of the new processes, but usually answer only at a single question and for very selected patients.

For this reason, the SIRIC Montpellier Cancer proposes to develop a prospective and regional Clinical Database Project and regional biological collection (blood and tumor samples), which is an expanding data collection designed to contribute to a better understand the patient's management with brain metastases including quality of life and neuropsychological/cognitive aspects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years
2. Radiological diagnosis of brain metastases
3. Patient eligible for neurosurgical exeresis or treatment by radio-surgery
4. Patient treated in a neurosurgery center of the Languedoc-Roussillon region (whatever therapeutic treatment realized on primary tumor)
5. Present brain metastases not previously treated
6. Signed informed consent
7. Patient affiliated to a national insurance system or beneficiary of such a system

Exclusion Criteria:

1. Patient with primary brain tumor
2. Impossibility to be regularly monitored for psychological, family, social, or geographical reasons
3. Subject under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who had a histological study of their brain metastases | 24 months
Number of patients who had a neurosurgery of their brain metastases | 24 months
Number of patients who had a radiotherapy of their brain metastases | 24 months
Number of patients who had a chemotherapy of their brain metastases | 24 months

SECONDARY OUTCOMES:
Quality of life by using the quality of life questionnaire core (QLQ-C30). | 24 months
  The EORTC QLQ-C30 uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Quality of life by using the quality of life questionnaire - brain neoplasm (BN20) | 24 months
  The QLQ-BN20 questionnaire contains 20 items organized into four scales; future uncertainty (3 items), visual disorder (3 items); motor dysfunction (3 items); and communication deficit (3 items), and seven single items (headaches, seizures, drowsiness, hair loss, itchy skin, weakness of legs, and bladder control). All items are rated on a four-point Likert-type scale ('1=not at all', 2='a little', '3=quite a bit' and '4=very much'), and are linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Cognitive and neuropsychological functions by using Montreal Cognitive assessment (MoCA) | 24 months
  Performance on the MoCA (Range : 0-30; higher score indicates better performance)
Overall Survival | Approximately 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Luc Bauchet, MD, Principal Investigator — Centre hospitalier de Montpellier
Locations (12):
- France (12):
  - Centre hospitalier régional et universitaire de Nîmes, Nîmes, Gard
  - Centre médical Oncogard, Nîmes, Gard
  - Clinique les Franciscaines, Nîmes, Gard
  - Laboratoire d'anatomo-pathologie de Nîmes, Nîmes, Gard
  - Centre médical Oncodoc Béziers, Béziers, Hérault
  - Centre d'Anatomie et Cytologie Pathologiques de Grabels, Grabels, Hérault
  - Centre hospitalier régional et universitaire de Montpellier, Montpellier, Hérault
  - Clinique Clémentville, Montpellier, Hérault
  - Clinique du Millénaire, Montpellier, Hérault
  - Institut régional du cancer, Montpellier, Hérault
  - Centre hospitalier de Perpignan, Perpignan, Pyrénées-orientales
  - Clinique Saint-Pierre, Perpignan, Pyrénées-orientales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis FG, Dolecek TA, McCarthy BJ, Villano JL. Toward determining the lifetime occurrence of metastatic brain tumors estimated from 2007 United States cancer incidence data. Neuro Oncol. 2012 Sep;14(9):1171-7. doi: 10.1093/neuonc/nos152. Epub 2012 Aug 16. PMID 22898372
- [Background] Fox BD, Cheung VJ, Patel AJ, Suki D, Rao G. Epidemiology of metastatic brain tumors. Neurosurg Clin N Am. 2011 Jan;22(1):1-6, v. doi: 10.1016/j.nec.2010.08.007. PMID 21109143
- [Background] Smedby KE, Brandt L, Backlund ML, Blomqvist P. Brain metastases admissions in Sweden between 1987 and 2006. Br J Cancer. 2009 Dec 1;101(11):1919-24. doi: 10.1038/sj.bjc.6605373. Epub 2009 Oct 13. PMID 19826419
- [Background] Kocher M, Soffietti R, Abacioglu U, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Collette S, Collette L, Mueller RP. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. J Clin Oncol. 2011 Jan 10;29(2):134-41. doi: 10.1200/JCO.2010.30.1655. Epub 2010 Nov 1. PMID 21041710